CLINICAL TRIAL: NCT04774198
Title: Perioperative Immune Function and Clinical Complications in Pancreaduodenectomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, Clinical Professor, Rigshospitalet, Denmark
Other Study IDs: H-17024315
Record Dates: First submitted 2021-01-31; First posted 2021-03-01 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Full blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Occurrence of persistent postoperative hypotension: Patients with need for noradrenaline the morning after surgery to maintain middle arterial blood-pressure (MAP)>65 mmHg, after pancreaticoduodenectomy.
  Interventions: Diagnostic Test: blood sample
- No occurrence of persistent postoperative hypotension: Patients without need for noradrenaline the morning after surgery to maintain middle arterial blood-pressure (MAP)>65 mmHg, after pancreaticoduodenectomy.
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample — Blood samples are collected within 24 hours before the surgical procedure, on postoperative day two and seven. Samples collected are as following: TruCulture, flow cytometry, markers of systemic inflammation (Plasma level of pro- and anti-inflammatory molecules assed by Olink inflammation panel, leucocytes, differential count, hemoglobin, thrombocytes and CRP)

SUMMARY:
Perioperative immunologic signatures can predict the risk of postoperative complications.

The results will be puplished as two smanuscripts. The manuscript will focus on preoperative immunologisk data,the second manuscript will include both pre- and postoperative data.

DETAILED DESCRIPTION:
OBJECTIVE Establish evidence for perioperative immunologic risk stratification of patient's risk for clinically postoperative inflammatory complications as a basis for future mechanism-based intervention studies.

Combining detailed immune assessment from cell-receptors to cell expression, cytokines, and complications with a temporal aspect is innovative and provides highly warranted novel multidimensional immunological insight.

METHODS Adult patients scheduled for PD on the suspicion of pancreatic cancer excluding patients receiving immunomodulating treatment 1 month properatively and/or autoimmune diseases. Patients scheduled for simultaneous procedures on major blood vessels, and/or adjacent organs (spleen, liver) are also not included. Inoperable patients, for instance, due to carcinosis, circulatory/ventilatory instability hindering procedure completion and/or concomitant surgery on major blood vessels, spleen, or liver, are excluded post-inclusion and will not be part of the primary analysis. Patients eligible for inclusion will be identified before their appointment at the Gastrosurgical Dept., Rigshospitalet which is the largest DK and North-European center with about 200 PD/yr annually.

Primary outcome:

Persistent postoperative hypotension, defined as need for vassopressor infussion on the morning after surgery to maintain middle arterial bloodpressure >65 mmHg

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for PD on the suspicion of pancreatic cancer
* Patients able to follow standardised surgical procedure including TIVA anaesthesia with epidural

Exclusion Criteria:

* Bilirubin >100 µmol/ltr
* Patients receiving immunomodulating treatment 1 month properatively and/or autoimmune diseases and patients non-cenacerous cystic lessions
* Patients scheduled for simultaneous procedures on major arterial blood vessels, and/or adjacent organs (spleen, liver)
* Inoperable patients, for instance, due to carcinosis, circulatory/ventilatory instability hindering procedure completion and/or concomitant surgery on major arterial blood vessels, spleen, or liver, are excluded post-inclusion and will not be part of the primary analysis
* ongoing treatment with glucocortocoid, anti-tnf-alpha etc.
* patients diagnosed with rheumatological diseases, IBD or chronic infection (eg. HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for PD on the suspicion of pancreatic cancer excluding patients receiving immunomodulating treatment 1 month properatively and/or autoimmune diseases and patients non-cenacerous cystic lessions. Patients scheduled for simultaneous procedures on major arterial blood vessels, and/or adjacent organs (spleen, liver) are also not included. Inoperable patients, for instance, due to carcinosis, circulatory/ventilatory instability hindering procedure completion and/or concomitant surgery on major arterial blood vessels, spleen, or liver, are excluded post-inclusion and will not be part of the primary analysis. Patients eligible for inclusion will be identified before their appointment.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with persistent postoperative hypotension (<65 mmHg) after surgery | 24 hours
  Need for vasopressor infusion (noradrenaline) to maintain middle arterial blood pressure >65 mmHg, the morning after pancreaticoduodenectomy.

SECONDARY OUTCOMES:
Number of patients with infection | 30 days
  Ex. surgical site infection, pneumonia, sepsis, etc, based upon international criteria (eg. center for disease control)
Number of patients with occurrence (yes/no) of systemic inflammatory response syndrome (SIRS) at any time during the first 30 days | 30 days
  SIRS defined as two or more of either of the following four criteria: i) temperature <36°C or >38°C, ii) heart rate >90/min., iii) respiratory rate >20/min and/or iv) white blood cell count (WBC) <4x109/L (<4000/mm³), >12x109/L (>12,000/mm³) or ≥10% bands neutrophils.
Number of patients with severe clinical intra- and postoperatove complications | 30 days
  Complications assessed by Clavien-Dindo classification and Comprehensive Clinical complication Index (CCI) ( (i.e. anastomotic leakage, reoperation, thrombosis, bleeding, etc.)
Number of patients with severe clinical intra- and postoperative complications | 30 days
  Complications assessed by SOFA score including single organ system deviation
Number of patients with severe perioperative physiological deviations | 30 days
  Frequency og physiological deviation Monitored by WARD-clinical support system (i.e hypotension, desaturation, tachycardia, etc.).
Number of patients with development of delirium after surgery | 7 days
  Development of delirium measured with the 3D-CAM score

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, DMSci, Study Chair — Rigshospitalet, Denmark; Sisse R Ostrowski, DMSci, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided